CLINICAL TRIAL: NCT00971113
Title: Impact of a Jelly Containing Short Chain Fructo-oligosaccharides and Sideritis Euboea Extract on Human Gut Microflora
Brief Title: Prebiotic Effect of a Jelly Containing Short Chain Fructo-Oligosaccharides and Sideritis Euboea Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: Hellenic Republic Ministry of Development (Unknown); Jotis S.A. Food Industry (Unknown)
Responsible Party: Kyriacou Adamantini, Lecturer, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 05PAV 363
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sc-FOS+Sideritis euboea group (Experimental): Jelly supplemented with short chain fructooligosaccharides and Sideritis euboea extract
  Interventions: Dietary Supplement: sc-FOS and Sideritis euboea extract
- placebo group (Placebo Comparator): Jelly without short-chain fructooligosaccharides and Sideritis euboea
  Interventions: Dietary Supplement: sc-FOS and Sideritis euboea extract

INTERVENTIONS:
Dietary Supplement: sc-FOS and Sideritis euboea extract — dietary supplement: jelly with 5g sc-FOS and 0.3g Sideritis euboea extract per daily portion for 30 days
  placebo food: jelly with no sc-FOS and Sideritis euboea

SUMMARY:
The human intestinal microflora is characterized as a complex and dynamic microbial ecosystem with crucial contribution to our nutrition and welfare. Health-promoting genera such as Bifidobacterium spp. and Lactobacillus spp. play a key role in digestion of nutrients, production of short chain fatty acids and vitamins, inhibition of harmful bacteria, immunostimulation, reduction of blood cholesterol and ammonia levels and restoration of normal flora after antibiotic therapy. Proteolytic species such as toxin-producing clostridia and toxigenic E. coli are considered as potential pathogens with detrimental effects to human host.

Recently, part of novel food research is directing towards the concept of prebiotics e.g. food ingredients that are not hydrolyzed by the human gastrointestinal tract and beneficially affect the host by selectively stimulating the growth and/or activity of one or limited number of bacteria in the colon that can improve host health.

Fructo-oligosaccharides and inulin, are considered as the most extensively studied and well-established prebiotics. In vitro and in vivo data suggest the bifidogenic effect of inulin and oligofructose, which can be attributed to their selective fermentation by Bifidobacterium species. Due to their documented prebiotic properties, both inulin and FOS are increasingly applied in novel food product development through the fortification of commonly ingested foodstuffs.

The aim of this study is to evaluate the in vivo prebiotic effect of a functional food containing short-chain fructo-oligosaccharides (sc-FOS) and Sideritis euboea extract on the faecal microflora composition of healthy human volunteers.

DETAILED DESCRIPTION:
In this randomized, double-blinded, placebo-controlled clinical study we aimed to evaluate the in vivo prebiotic effects of a functional food containing short-chain fructo-oligosaccharides (sc-FOS) and Sideritis euboea extract on human faecal microflora. Sixty-four healthy volunteers (26 men and 38 women) (age range:22-51) were assigned to consume daily a jelly containing 5 g sc-FOS and 0.3 g S.euboea extract or a placebo for 30 d. Stool samples were collected prior to the study on day 15 and 30 of intervention and 2 weeks after. Enumeration of faecal bacteria was performed by plate count techniques. Gastrointestinal side effects were recorded during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects

Exclusion Criteria:

* History of gastrointestinal disease
* Chronic diseases (i.e.,diabetes,cardiovascular diseases, hyperlipidemia, autoimmune disorders)
* History of epileptic seizures
* Extreme dietary behaviours
* Consumption of antibiotics and other medication 2 months prior and during the investigation period

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
to evaluate the in vivo prebiotic effect of an jelly containing sc-FOS and Sideritis euboea extract on the faecal microflora composition and to evaluate the effect of jelly containing sc-FOS and Sideritis euboea extract on gastrointestinal symptoms | 30d intervention and 2 wks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Adamantini Kyriacou, Ass. Professor, Study Director — Harokopio University
Locations (1):
- Harokopio University, Kallithea, Attica, Greece